CLINICAL TRIAL: NCT03926026
Title: A Multi-Center, Randomized, Double-Masked, Placebo-Controlled, Dose-Escalation, Phase 2 Study Evaluating the Safety and Tolerability of NCX 4251 (Fluticasone Propionate Nanocrystal) Ophthalmic Suspension, 0.1% QD and BID for the Treatment of Acute Exacerbations of Blepharitis
Brief Title: Study Evaluating the Safety and Tolerability of NCX 4251 for the Treatment of Acute Exacerbations of Blepharitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nicox Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCX-4251-01
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Fluticasone

STUDY DESIGN:
Intervention Model Description: sequential dose-escalating cohorts -- Cohort 1 (2 parallel groups) and Cohort 2 (2 parallel groups)
Who Masked: Participant, Investigator
Masking Description: double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NCX 4251 QD (Experimental): NCX 4251 Ophthalmic Suspension, 0.1% once daily for 14 days
  Interventions: Drug: Fluticasone Propionate
- Placebo QD (Placebo Comparator): Placebo once daily for 14 days
  Interventions: Drug: Placebo
- NCX 4251 BID (Experimental): NCX 4251 Ophthalmic Suspension, 0.1% twice daily for 14 days
  Interventions: Drug: Fluticasone Propionate
- Placebo BID (Placebo Comparator): Placebo twice daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone Propionate — NCX 4251 Ophthalmic Suspension, 0.1%
  Other Names: NCX 4251
  Arms: NCX 4251 BID; NCX 4251 QD
Drug: Placebo — NCX 4251 Ophthalmic Suspension, 0%
  Arms: Placebo BID; Placebo QD

SUMMARY:
This is a multi-center, randomized, double-masked, placebo-controlled, Phase 2 study evaluating the safety and tolerability of NCX 4251 (fluticasone propionate nanocrystal) Ophthalmic Suspension 0.1% QD and BID for the treatment of acute exacerbations of blepharitis. The study will be performed in two sequential dose escalating cohorts.

The study is designed to select the dose(s) of NCX 4251 to advance into the next stage of development, and to assess the safety and tolerability of NCX 4251 Ophthalmic Suspension.

ELIGIBILITY:
Inclusion Criteria:

* history of blepharitis and meet qualifying criteria for an acute exacerbation of blepharitis in both eyes at Screening and Baseline/Day 1 Visits
* have a qualifying best-corrected visual acuity

Exclusion Criteria:

* abnormality of the eyelids or lashes (other than blepharitis), or previous eyelid surgery
* IOP > 21 mmHg at Screening or Baseline/Day 1 Visits
* use of steroids in the past 30 days or retinoids in the past 12 months
* uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicox Ophthalmics, Study Director — Nicox Ophthalmics, Inc.
Locations (1):
- Texan Eye, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NCX 4251 QD -- Cohort 1: NCX 4251 Ophthalmic Suspension, 0.1% once daily for 14 days
  Fluticasone Propionate: NCX 4251 Ophthalmic Suspension, 0.1%
- Placebo QD -- Cohort 1: Placebo once daily for 14 days
  Placebo: NCX 4251 Ophthalmic Suspension, 0%
- NCX 4251 BID -- Cohort 2: NCX 4251 Ophthalmic Suspension, 0.1% twice daily for 14 days
  Fluticasone Propionate: NCX 4251 Ophthalmic Suspension, 0.1%
- Placebo BID -- Cohort 2: Placebo twice daily for 14 days
  Placebo: NCX 4251 Ophthalmic Suspension, 0%
Period: Overall Study
Arm/Group | NCX 4251 QD -- Cohort 1 | Placebo QD -- Cohort 1 | NCX 4251 BID -- Cohort 2 | Placebo BID -- Cohort 2
Started | 10 | 5 | 10 | 11
Completed | 10 | 5 | 10 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The primary outcome measure was based on the study eye
Units Other Than Participants: study eyes
Groups:
- NCX 4251 QD (Cohort 1): NCX 4251 Ophthalmic Suspension, 0.1% once daily for 14 days
  Fluticasone Propionate: NCX 4251 Ophthalmic Suspension, 0.1%
- Placebo QD (Cohort 1): Placebo once daily for 14 days
  Placebo: NCX 4251 Ophthalmic Suspension, 0%
- NCX 4251 QD (Cohort 2): NCX 4251 Ophthalmic Suspension, 0.1% twice daily for 14 days
  Fluticasone Propionate: NCX 4251 Ophthalmic Suspension, 0.1%
- Placebo QD (Cohort 2): Placebo twice daily for 14 days
  Placebo: NCX 4251 Ophthalmic Suspension, 0%
- Total: Total of all reporting groups
Arm/Group | NCX 4251 QD (Cohort 1) | Placebo QD (Cohort 1) | NCX 4251 QD (Cohort 2) | Placebo QD (Cohort 2) | Total
Number analyzed (Participants) | 10 | 5 | 10 | 11 | 36
Number analyzed (study eyes) | 10 | 5 | 10 | 11 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5 | 5 | 15
  >=65 years | 6 | 4 | 5 | 6 | 21
Age, Continuous [Mean (Full Range); unit: years] | 63.5 [28 to 84] | 67.8 [48 to 88] | 58.3 [28 to 84] | 64.5 [48 to 78] | 65.4 [28 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 7 | 5 | 21
  Male | 3 | 3 | 3 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 9 | 5 | 9 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 10 | 5 | 9 | 11 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 10 | 11 | 36
Composite score of eyelid discomfort, eyelid margin redness, and debris [Mean (Full Range); unit: units on a scale] — Eyelid margin discomfort (0=none to 3=severe) + eyelid margin redness (0=none/normal to 3=severe) + debris (0=none to 3=severe) for a composite total score ranging from 0 to 9.
  Eyelid margin discomfort reported by the participant; eyelid margin redness and eyelid debris evaluated by the investigator at the slit lamp.
  units on a scale | 4.7 [4 to 6] | 5 [4 to 7] | 4.6 [4 to 6] | 4.5 [3 to 6] | 4.8 [3 to 7]

OUTCOME MEASURES:

1. Primary Outcome: COHORT 1 and 2 COMBINED: Mean Change From Baseline to Day 14 in the Composite (Sum) Score of Signs & Symptoms of Blepharitis
Description: COHORT 1 and 2 COMBINED: Mean change from baseline in Composite (Sum) Score of Eyelid Margin Redness (0=none to 3=severe scale), Eyelid Debris (0=none to 3=severe scale), and Eyelid Discomfort (0=none to 3=severe scale)
Time Frame: 14 days
Population: intent-to-treat population
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: study eyes
Groups:
- NCX 4251 (Cohort 1 & 2 Combined): NCX 4251 Ophthalmic Suspension, 0.1% once or twice daily for 14 days
  Fluticasone Propionate: NCX 4251 Ophthalmic Suspension, 0.1%
- Placebo (Cohort 1 & 2 Combined): Placebo once or twice daily for 14 days
  Placebo: NCX 4251 Ophthalmic Suspension, 0%
Arm/Group | NCX 4251 (Cohort 1 & 2 Combined) | Placebo (Cohort 1 & 2 Combined)
Number analyzed (Participants) | 20 | 16
Number analyzed (study eyes) | 20 | 16
units on a scale | -2.0 [-4 to 1] | -1.2 [-2 to 1]
Statistical Analysis 1: Comparison: NCX 4251 (Cohort 1 & 2 Combined) vs Placebo (Cohort 1 & 2 Combined); Test type: Superiority; p = 0.0471, t-test, 2 sided; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.5 to 0]

2. Secondary Outcome: COHORT 2: Mean Change From Baseline to Day 14 in the Composite (Sum) Score of Signs & Symptoms of Blepharitis
Description: COHORT 2: Mean change from baseline in Composite (Sum) Score of Eyelid Margin Redness (0=none to 3=severe scale), Eyelid Debris (0=none to 3=severe scale), and Eyelid Discomfort (0=none to 3=severe scale)
Time Frame: 14 days
Population: intent-to-treat population
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: study eyes
Groups:
- NCX 4251 BID (Cohort 2): NCX 4251 Ophthalmic Suspension, 0.1% twice daily for 14 days
  Fluticasone Propionate: NCX 4251 Ophthalmic Suspension, 0.1%
- Placebo BID (Cohort 2): Placebo twice daily for 14 days
  Placebo: NCX 4251 Ophthalmic Suspension, 0%
Arm/Group | NCX 4251 BID (Cohort 2) | Placebo BID (Cohort 2)
Number analyzed (Participants) | 10 | 11
Number analyzed (study eyes) | 10 | 11
units on a scale | -1.7 [-3 to -1] | -1.1 [-2 to 1]

3. Secondary Outcome: COHORT 1: Mean Change From Baseline to Day 14 in the Composite (Sum) Score of Signs & Symptoms of Blepharitis
Description: COHORT 1: Mean change from baseline in Composite (Sum) Score of Eyelid Margin Redness (0=none to 3=severe scale), Eyelid Debris (0=none to 3=severe scale), and Eyelid Discomfort (0=none to 3=severe scale)
Time Frame: 14 days
Population: intent-to-treat population
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: study eyes
Arm/Group | NCX 4251 QD (Cohort 1) | Placebo QD (Cohort 1)
Number analyzed (Participants) | 10 | 5
Number analyzed (study eyes) | 10 | 5
units on a scale | -2.2 [-4 to 1] | -1.2 [-2 to 0]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | NCX 4251 QD | Placebo QD | NCX 4251 BID | Placebo BID
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 0/5 | 5/10 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NCX 4251 QD (N=10) | Placebo QD (N=5) | NCX 4251 BID (N=10) | Placebo BID (N=11)
eyelid margin crusting (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
conjunctival hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
instillation site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT03926026/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT03926026/SAP_001.pdf